CLINICAL TRIAL: NCT04880174
Title: SARS-COV-2 Seroprevalence and Seroconversion Among Employees of the Universitair Ziekenhuis Brussel Following mRNA COVID-19 Vaccination
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVEMUZ-2
Record Dates: First submitted 2021-04-16; First posted 2021-05-10 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: SARS-CoV Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- General arm (Other): All patients follow this arm. Patients will undergo 3 blood sample testings at 3 different time points and have to fill in a questionnaire at 3 different time points
  Interventions: Diagnostic Test: serological testing

INTERVENTIONS:
Diagnostic Test: serological testing — Antibody testing for Sars-COV-2 antibodies in blood.

SUMMARY:
A novel zoonotic coronavirus was discovered in Wuhan (Hubei Province, China) mid-December 2019 and was named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The virus rapidly spread to the rest of the world, including Europe and explicitly affects the respiratory system, generating Coronavirus disease 2019 (COVID-19).

This study is a monocentric interventional prospective and retrospective cohort study. After signing a written informed consent, participants will be recruited for questionnaire completion and blood sampling. Sample storage and analysis will be performed at the laboratory of microbiology of the UZ Brussel.

To document SARS-CoV-2 seroprevalence and seroconversion among employees of the UZ Brussel after mRNA vaccination for SARS-CoV-2, namely at 8 weeks after first vaccination, 6 months after first vaccination and 12 months after first vaccination.

DETAILED DESCRIPTION:
A novel zoonotic coronavirus was discovered in Wuhan (Hubei Province, China) mid-December 2019 and was named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The virus rapidly spread to the rest of the world, including Europe and explicitly affects the respiratory system, generating Coronavirus disease 2019 (COVID-19).

UZ Brussel employees presenting symptoms suggestive of COVID-19 are offered to be tested with real-time PCR on nasopharyngeal swabs. As asymptomatic infections have been described and as the PCR can be negative when taken late after onset of symptoms, serologic tests can be performed. The SARS-CoV 2003 epidemic demonstrated that serological assays were a useful diagnostic tool of non-acute infections. Although it is still uncertain whether convalescing patients have a risk of re-infection, recent data suggest that SARS-CoV-2 antibodies could protect at least for some time from subsequent viral exposures.

As the COVID-19 pandemic had devastating medical, economic and social consequences, safe and effective prophylactic vaccines were urgently needed. And thus several candidate vaccines against SARS-CoV-2 have been developed. During the first weeks of the vaccination campaign, the health care workers of the UZ Brussel, were invited to receive the BNT162b2 (Pfizer) vaccine.

Consequently, the investigators aim to prospectively document the SARS-CoV-2 seroprevalence and seroconversion among vaccinated employees of the UZ Brussel, at three different time points, namely 6 weeks (+/- 2 weeks; T1), 6 months (+/- 1 month; T2) and 12 months (+/- 1 month; T3) after the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Any adult employee of the UZ Brussel at T1 who has been vaccinated at the UZ Brussel with mRNA COVID-19 vaccine (Comirnaty®) between the 19th of January and the 5th of February 2021 after participating to phase 4 of the COVEMUZ study (with a maximum of 5 days difference between blood drawel and vaccination) and has provided a signed informed consent.

Exclusion Criteria:

* UZ Brussel employees not active during the inclusion period (T1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
seroprevalence | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To document SARS-CoV-2 seroprevalence among employees of the UZ Brussel after mRNA vaccination for SARS-CoV-2, at 8 (+/- 2) weeks after the first vaccination (T1); and 6 and 12 months after the first vaccination (T2 and T3) using a validated immuno-assay for detection of SARS-CoV-2 IgG antibodies
Seroconversion | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To document SARS-CoV-2 seroconversion among employees of the UZ Brussel after mRNA vaccination for SARS-CoV-2, at 8 (+/- 2) weeks after the first vaccination (T1); and 6 and 12 months after the first vaccination (T2 and T3) using a validated immuno-assay for detection of SARS-CoV-2 IgG antibodies

SECONDARY OUTCOMES:
SARS-CoV-2 seroprevalence before and after vaccination | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To compare the SARS-CoV-2 seroprevalence before vaccination with the SARS-CoV-2 prevalence after vaccination among employees of the UZ Brussel.
incidence of new definite cases | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To document the incidence of new definite cases of COVID-19 (based on self-reported positive PCR testing on nasopharyngeal swab) among vaccinated employees of the UZ Brussel over a period of a year.
incidence of new probable cases | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To document the incidence of new probable cases of COVID-19 (based on the study questionnaire filled in by the participants) among vaccinated employees of the UZ Brussel over a period of a year.
antibody kinetics and antibody neutralisation capacity | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To document the SARS-CoV-2 antibody kinetics and antibody neutralisation capacity after vaccination.
antigen-specificity of the SARS-CoV-2-specific T cells | Change from baseline to 8 weeks, 6 months and 12 months timepoint
  To determine the antigen-specificity of the SARS-CoV-2-specific T cells as well as their phenotype and functionality.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No